CLINICAL TRIAL: NCT04834700
Title: Comparison of Hands-on Versus Online Learning in Teaching Ultrasound Skills for Eye
Brief Title: Comparison of Hands-on Versus Online Learning About Ocular Ultrasound
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-09-174
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-03

CONDITIONS: Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hands-on group (No Intervention): The doctors who participated in the study will be educated ocular ultrasound scanning method by hands-on about 20 minutes, and perform ocular ultrasound scans on two standard patients.
- online group (Other): The doctors who participated in the study will be educated ocular ultrasound scanning method by online lecture about 20 minutes, and perform ocular ultrasound scans on two standard patients.
  Interventions: Other: online group

INTERVENTIONS:
Other: online group — In terms of teaching ultrasound, video lectures will be conducted rather than hands-on, which is the traditional method.
  Arms: online group

SUMMARY:
In patients who visit an emergency room with ocular symptoms, point-of-care ultrasound can quickly identify several emergency diseases. While training of eye ultrasound skills is useful for emergency physicians, hands-on education is risky in pandemic situation such as coronavirus disease 19 (COVID19). As a solution to this, non-face-to-face education via online has been on the rise. The investigators hypothesized that even an online education is enough to perform basic eye ultrasound by emergency physician.

DETAILED DESCRIPTION:
Since the eye is an superficial organ, it has excellent access to ultrasound. Also, the eye has a liquid-filled structure (vitreous body), it is suitable for obtaining some important findings with bedside ultrasound. In patients who visit an emergency room with ocular symptoms, point-of-care ultrasound can quickly identify several emergency diseases. While training of eye ultrasound skills is useful for emergency physicians, hands-on education is risky in pandemic situation such as COVID19. As a solution to this, non-face-to-face education via online has been on the rise. The investigators hypothesized that even an online education is enough to perform basic eye ultrasound by emergency physician.

ELIGIBILITY:
Inclusion Criteria for doctors:

* Those who have received basic ultrasound education but have not received ocular ultrasound education
* Residents and interns working in the emergency room
* Those who voluntarily agree to participate in the research through the recruitment announcement

Inclusion Criteria for standard patients:

* Adults over 18 years of age without eye-related symptoms
* Those who do not have unusual findings in the eye when scanning by ultrasound
* Those who voluntarily agree to participate in the research through the recruitment announcement

Exclusion Criteria for standard patients:

* Those with a history of ophthalmic diseases
* Those who have a history of ophthalmic surgery such as lens implantation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
scan score | through study completion, an average of 1 year
  We make our own guideline to evaluate ocular ultrasound scans. The ocular ultrasound images performed participants are evaluated according to the guideline.
  We compare the scores of the hands-on group and the online group to see if there is a significant difference between the two groups.

SECONDARY OUTCOMES:
Optic nerve sheath diameter (ONSD) | through study completion, an average of 1 year
  Two ultrasound experts measure the standard patient's ONSD and use it as a reference value.
  The course of ocular ultrasound scanning involves measuring ONSD. We compare the measured ONSD of the hands-on group and the online group to see if there is a significant difference between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Yoon, MD., PhD., Study Director — Samsung medical center, Emergency department
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No